CLINICAL TRIAL: NCT06413953
Title: A Phase I Clinical Study of Tolerability and Pharmacokinetics of TQB3107 Tablets in Patients With Malignant Tumors
Brief Title: A Clinical Study of TQB3107 Tablets in Patients With Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3107-I-01
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-12

CONDITIONS: Advanced Cancers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3107 tablets (Experimental): Dosing regimen 1 (20/28): 28 days per cycle (4 weeks), the medication is administered once daily for 5 consecutive days per week, followed by a 2-day break. The initial dose is a single fasting dose of C0, with a subsequent 7-day observation period.
  Dosing regimen 2 (28/28): 28 days per cycle, the medication is administered once daily for the entire 28-day period, all other dosing requirements are consistent with Regimen 1.
  Interventions: Drug: TQB3107 Tablets

INTERVENTIONS:
Drug: TQB3107 Tablets — TQB3107 tablets is protein inhibitor that inhibit tumor cell proliferation, and induce apoptosis, thereby exerting anti-tumor effects.

SUMMARY:
TQB3107 is a protein inhibitor that induces apoptosis and inhibits the proliferation of various tumor cells. This clinical study aims to evaluate the safety and tolerability of TQB3107 tablets in subjects with advanced malignancies, to determine the dose-limiting toxicities (DLTs), maximum tolerated dose (MTD) (if any), and the recommended dose for Phase II (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age≤ 75 years (calculated from the date of signing the informed consent); Score 0~1 point, estimated survival ≥ 3 months；
* Malignant tumors with no standard treatment regimen or disease progression or intolerance after prior standard therapy；
* The major organs are functioning well；
* Negative serum pregnancy test within 7 days prior to the first dose and must be a non-lactating subject, female and male subjects of childbearing potential should agree to use contraception throughout the study and for 6 months after the study ends;
* Subjects voluntarily participated in this study, signing the informed consent form and demonstrating good compliance.

Exclusion Criteria:

* Hematologic malignancy has or is suspected to involve the central nervous system, or primary central nervous system lymphoma;
* Received any anti-cancer therapy such as major surgery, chemotherapy and/or radiotherapy, immunotherapy, or targeted therapy within 4 weeks prior to the first dose;
* Combined with severe or not well-controlled diseases, which the investigator judges to be at greater risk of entering this study；
* Those with a history of drug addiction or substance abuse；
* Based on the investigator's judgement, subjects with concomitant diseases that pose a significant risk to their safety or compromise the study's completion, or subjects deemed unsuitable for enrollment due to other reasons, will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  DLT refers to toxicities that are associated with the drug and occur from the first medication administration to the end of the first treatment cycle, as defined by the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 toxicity assessment criteria.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 28 days)
  MTD is defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Phase II Recommended Dose (RP2D) | Baseline up to 24 months
  The recommended dose, determined after initial dose escalation and toxicity assessment, it is used to further evaluate the efficacy and safety of the drug.

SECONDARY OUTCOMES:
Elimination half-life (t1/2) | Day 1 of cycles 0 and 2: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; Days 1, 8 and 15 of cycle 1: in 30 minutes (pre-dose); Day 26 of cycle 1: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
  The time it takes for the concentration of the drug in the plasma to be reduced by 50%.
Time to Peak (Tmax) | Day 1 of cycles 0 and 2: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose；Days 1, 8 and 15 of cycle 1: in 30 minutes (pre-dose); Day 26 of cycle 1: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
  The time it takes to reach peak concentrations after administration.
Peak Concentration (Cmax) | Day 1 of cycles 0 and 2: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; Days 1, 8 and 15 of cycle 1: in 30 minutes (pre-dose); Day 26 of cycle 1: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
  Maximum plasma concentration of drug.
Area under the plasma concentration-time curve (AUC0-last) | Day 1 of cycles 0 and 2: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; Days 1, 8 15 of cycle 1: in 30 minutes (pre-dose); Day 26 of cycle 1: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
  The area enclosed by the plasma concentration curve against the timeline.
Steady-state peak concentration (Css-max) | Day 1 of cycle 0 and 2: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; Days 1, 8 and 15 of cycle 1: in 30 minutes (pre-dose); Day 26 of cycle 1: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
  The highest plasma drug concentration that occurs after stabilization.
Steady-state trough concentration (Css-min) | Day 1 of cycles 0 and 2: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; Days 1, 8 and 15 of cycle 1: in 30 minutes (pre-dose); Day 26 of cycle 1: in 30 minutes (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
  Minimum plasma drug concentration during dosing.
Objective Response Rate (ORR) | Up to 2 years
  The percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
Disease Control Rate (DCR) | Up to 2 years
  Proportion of patients whose tumors achieve remission (PR+CR) and stable disease (SD) after treatment and can maintain the minimum timeframe required according to accepted response evaluation criteria (e.g., RECIST version 1.1 for solid tumors).
Duration of Response (DOR) | Up to 2 years
  The time from first documented response to documented disease progression.
Progression-free survival (PFS) | Up to 2 years
  The time from the start of treatment to tumor progression or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 2 years
  The time from the start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Cen, Guangzhou, Guangdong, China